CLINICAL TRIAL: NCT06794021
Title: A One Week Randomized, Double Blind, Placebo Controlled, Clinical Study to Examine the Benefits of an Oral Product in Subjects With Menopausal Symptoms Including Vasomotor Symptoms (VMS).
Brief Title: One Week Clinical Study in Subjects With Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olly, PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UNLV20241205
Record Dates: First submitted 2025-01-06; First posted 2025-01-27 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Menopause
MeSH Terms: interventions — Dietary Supplements; gamma-Aminobutyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Oral dietary supplement. Instructions: Take 1 capsule when having a hot flash at the onset of a hot flash (not to exceed 1 capsule/day). Only treat 1 hot flash during a 24-hour period.
  Interventions: Other: Placebo
- Dietary Supplement with Proprietary Herbal Extract Blend and GABA (Active Comparator): Oral dietary supplement. Instructions: Take 1 capsule when having a hot flash at the onset of a hot flash (not to exceed 1 capsule/day). Only treat 1 hot flash during a 24-hour period.
  Interventions: Dietary Supplement: Dietary Supplement with Proprietary Herbal Extract Blend and GABA

INTERVENTIONS:
Dietary Supplement: Dietary Supplement with Proprietary Herbal Extract Blend and GABA — Eligible subjects will receive active product to take daily for seven days
  Arms: Dietary Supplement with Proprietary Herbal Extract Blend and GABA
Other: Placebo — Eligible subjects will receive Placebo to take daily for seven days
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to Examine the Benefits of an Oral Product in Subjects With Menopausal Symptoms. The main questions it aims to answer are:

1. To assess the efficacy for improvement of menopausal vasomotor symptoms within 24 hours compared to placebo through Daily Diary and Mobile Application
2. To assess the efficacy for improvement of menopausal vasomotor symptoms hours compared to placebo through days 2-6 Daily Diary and Mobile Application
3. To assess the efficacy of the investigation product on stress/anxiety, mood swings, headaches compared to placebo through days 1-6 and with use of Daily Diary, Mobile Application and validated questionnaires (GCS, MENQOL).
4. To assess the efficacy of the investigation product on mood, stress and sleep at 7 days post treatment using validated questionnaires (PSQI, PSS, POMS)

ELIGIBILITY:
Inclusion Criteria:

* Healthy Females aged 40 to 65 years,
* Self-reporting menopausal symptoms (> 5 hot flushes per day) and have been present for a minimum of previous 60 days prior to baseline visit.
* Reporting a variable cycle length of > 7 days different from normal
* BMI 20-40 kg/m2
* Able to read, understand, and complete the study questionnaire and records.
* Able to understand the study procedures.
* Able to comply with all study requirements.
* Written informed consent to participate in the study.
* Willingness to actively participate in the study and to come to the scheduled visits.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Immune insufficiency
* Women of childbearing potential including those still having a menstrual cycle on a regular basis who are not perimenopausal, menopausal or post-menopausal.
* History of hysterectomy
* Women on hormone replacement therapy
* Use of systemic corticosteroids or immunosuppressant drugs.
* Other diseases or medications that might directly interfere in the study or put the subject's health under risk.
* Employees of the institute or the brand owner or the manufactures of the product
* Cardiovascular-, chronic liver-, thyroid or kidney diseases; a history of cancer; a disease or condition that could influence the participants' ability to follow the study protocol,
* Alcohol or drug abuse
* Use of hormonal contraceptives within the last 3 months
* Use of other menopause supplements
* BP ≥160/110 mmHg
* Oophorectomy or amenorrhea > two years. Note- Habitual medicine and supplement intake will be registered prior to inclusion in the study.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Daily Diary - 24hr | from enrollment to the end of study at seven days
  To assess changes in menopausal vasomotor symptoms scores within 24 hours compared to placebo through Daily Diary.
Mobile App - 24hr | from enrollment to the end of study at seven days
  To assess changes in menopausal vasomotor symptoms scores within 24 hours compared to placebo through Mobile Application.

SECONDARY OUTCOMES:
Daily Dairy - Days 1-6 | from enrollment to the end of study at seven days
  To assess changes in menopausal vasomotor symptoms, stress/anxiety, mood swings, and headaches scores compared to placebo through days 1-6
Mobile App - Days 1-6 | from enrollment to the end of study at seven days
  To assess changes in menopausal vasomotor symptoms, stress/anxiety, mood swings, and headaches scores compared to placebo through days 1-6
Green Climacteric Scale (GCS) - Days 1-6 | from enrollment to the end of study at seven days
  To assess changes in stress/anxiety, mood swings, and headaches scores compared to placebo through days 1-6
Menopause-Specific Quality of Life (MENQOL) - Days 1-6 | from enrollment to the end of study at seven days
  To assess changes in menopausal vasomotor symptoms, stress/anxiety, mood swings, and headaches scores compared to placebo through days 1-6

OTHER OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) - Day 7 | from enrollment to the end of study at seven days
  To assess changes on mood, stress and sleep scores at 7 days post treatment
Perceived Stress Scale (PSS) - Day 7 | from enrollment to the end of study at seven days
  To assess changes on mood, stress and sleep scores at 7 days post treatment
Profile of Mood States questionnaire (POMS) - Day 7 | from enrollment to the end of study at seven days
  To assess changes on mood, stress and sleep scores at 7 days post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided